CLINICAL TRIAL: NCT00409695
Title: Dose Finding Study of Thymoglobulin (ATG) in Patients With Steroid-Refractory Acute Graft Versus Host Disease (aGVHD)
Brief Title: Thymoglobulin (ATG) Dose Finding Study
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-0370
Record Dates: First submitted 2006-12-07; First posted 2006-12-11 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Graft vs Host Disease
Keywords: Acute Graft versus Host Disease; aGVHD; Blood And Marrow Transplantation; Thymoglobulin; ATG
MeSH Terms: conditions — Graft vs Host Disease | interventions — thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Dose Thymoglobulin (ATG) (Experimental): High Dose Thymoglobulin (ATG): 1.25mg/kg by vein every other day for 3 doses (total dose = 3.75mg/kg)
  Interventions: Drug: High Dose Thymoglobulin (ATG)
- Low Dose Thymoglobulin (ATG) (Experimental): Low Dose Thymoglobulin (ATG): 2.5 mg /kg by vein every other day for 3 doses (total dose = 7.5 mg/ kg).
  Interventions: Drug: Low Dose Thymoglobulin (ATG)

INTERVENTIONS:
Drug: Low Dose Thymoglobulin (ATG) — 2.5 mg /kg by vein every other day for 3 doses (total dose = 7.5 mg/ kg).
  Other Names: ATG; Antithymocyte Globulin
  Arms: Low Dose Thymoglobulin (ATG)
Drug: High Dose Thymoglobulin (ATG) — 1.25mg/kg by vein every other day for 3 doses (total dose = 3.75mg/kg)
  Other Names: ATG; Antithymocyte Globulin
  Arms: High Dose Thymoglobulin (ATG)

SUMMARY:
Primary Objective:

* To determine the response and toxicity rate at day 56 of two different dose levels of thymoglobulin (ATG) [anti-thymocyte globulin (rabbit)] as a treatment of steroid-refractory acute graft versus host disease (aGVHD).

Secondary Objectives:

* To evaluate the response rate at day 28.
* To evaluate the overall survival and non-relapse mortality at 6 months.
* To determine the toxicity profile of thymoglobulin when used for the treatment of steroid-refractory aGVHD in each of two dose schedules.
* To characterize the pharmacokinetic profile of thymoglobulin in each of two dose schedules.
* To analyze biomarkers of cellular drug effect by quantifying T-cell apoptosis in aims of finding the minimal effective dose.
* To determine immune-reconstitution after administration of thymoglobulin to patients with steroid-refractory aGVHD for each dose schedule.

DETAILED DESCRIPTION:
GvHD is a common side effect of a stem cell transplant. It is caused by a type of white blood cell (a lymphocyte). ATG is designed to kill lymphocytes and is commonly used to help prevent or treat GvHD and to treat steroid-refractory aGvHD.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will be asked questions about your medical history. You will have a complete physical exam. You will have blood drawn (about 2 tablespoons) for routine tests and to check for any viral infections. Women who are able to have children must have a negative blood (about 1 teaspoon) or urine pregnancy test. You will also have a biopsy of the site that is suspected to be affected by aGvHD. The study doctor will describe the type of biopsy procedure you will have, which will depend on the part of the body that is affected by the disease. If you had an earlier biopsy performed that confirmed aGvHD, you will not need a biopsy repeated for this study.

If you are found to be eligible to participate in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. Participants in Group 1 will receive a higher dose of ATG by vein. Participants in Group 2 will receive a lower dose of ATG by vein. You will have an equal chance of being in 1 of the 2 groups. Participants in both groups will receive doses of ATG over 4-6 hours, 1 time a day every other day for a total of 3 doses.

During this study, you will be able to remain on steroids and any other drugs you may be receiving for treatment of aGvHD (such as tacrolimus or cyclosporine). You will also have blood drawn (about 1 teaspoon) to learn the effect of ATG on the lymphocytes.

You will be taken off this study, if the disease is stable as determined by the study doctor, if the disease gets worse, or you experience any intolerable side effects. If you are taken off this study, your study doctor will discuss other treatment options with you.

After you finish receiving the study medication, you will come to the clinic at regularly scheduled follow-up visits. At first, you will be seen in the clinic once a week for 1 month. You will also have additional blood drawn (about 2 teaspoons) for biomarker testing (testing that looks at how the drug is working in your body). After the first month of follow-up visits, you will come in for visits every other week while you are on this study, which will continue until you have at least 2 consecutive (back to back) evaluations of the disease status to see if the disease is stable.

This is an investigational study. ATG is FDA approved and commercially available. You and/or your insurance provider will be financially responsible for the cost of ATG while you are on this study. Up to 40 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent their first allogeneic transplant for any malignancy and with any cell (bone marrow, peripheral stem cell, cord blood) or donor (matched or mismatched related or unrelated) source.
2. Biopsy-proven, grade II-IV aGVHD following allogeneic hematopoietic stem cell transplantation (HSCT) of any source (bone marrow, peripheral blood or cord blood stem cells). Enrollment may be started prior to results of biopsy in cases of high clinical suspicion for aGVHD.
3. Early steroid-refractory aGVHD. This is defined as any NR or PD after a minimum of 3 days and not more than 1 week of 1 mg/kg/day of methylprednisolone.
4. Ability to sign informed consent.
5. Ability to return for clinical follow-up as specified in the protocol.
6. Inability to taper as defined by patients on < or = 1 mg/kg/day of methylprednisolone but unable to further taper without resultant increase of acute GVHD stage.
7. Patients with a reflare of a GVHD defined as worsening of 1 stage of acute GVHD in a patient who initially responded.

Exclusion Criteria:

1. Relapsed malignancy.
2. Acute GVHD as a result of a second or subsequent transplant or donor lymphocyte infusion (DLI).
3. Active, uncontrolled infection.
4. Patients who have received any second-line of immunosuppressive treatment for GVHD beyond corticosteroids and calcineurin inhibitors. Topical steroids, oral budesonide and extracorporeal photochemotherapy started at the time of steroids are allowed.
5. Life-threatening infusion reaction or hypersensitivity to any formulation of ATG in the past.
6. Patients who are pregnant or are breast feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Response Rate | Day 56
  Response assessed at day 56, and a complete response or partial response considered a success. A toxic event defined as a life threatening infection, any death due to infection, or any death considered to be directly related to the administration of ATG.

CONTACTS AND LOCATIONS:
Overall Officials: Amin M. Alousi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States